CLINICAL TRIAL: NCT06022783
Title: The Effectiveness of Virtual Reality Intervention on Stress Levels of Surgical Nurses: A Crossover Designed Study
Brief Title: Effect of Virtual Reality Intervention on Stress Levels of Surgical Nurses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Seher Ünver, Associate Professor, Trakya University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2023-KAEK-655
Record Dates: First submitted 2023-08-24; First posted 2023-09-05 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Nurse; Stress; Virtual Reality
Keywords: surgical nurses; stress; virtual reality intervention

STUDY DESIGN:
Intervention Model Description: crossover designed randomized controlled study
Who Masked: Outcomes Assessor
Masking Description: The data analysed by a independent researcher from the data collection and coding procedures.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- with VR-G (Experimental): The nurses in this procedure were asked to watch a relaxing video with using VR-G for 20 minutes at their break time.
  Interventions: Other: Virtual reality intervention
- no VR-G (No Intervention): The nurses in this procedure did not watch any video and completed their routine working shift and break times.

INTERVENTIONS:
Other: Virtual reality intervention — Watching a relaxing video with using VR-G for 20 minutes
  Arms: with VR-G

SUMMARY:
The aim this crossover designed study is to examine the effect of watching a relaxing video with using virtual reality glasses (VR-G) during the break period of a working shift on the stress levels of surgical nurses.

Nurses will be asked to watch a relaxing video with using VR-G for 20 minutes at their break time (the first procedure).

After one-week wash-out period, researchers will compare second procedure (no video watch with VR-G) to see if there is any difference on the stress levels of the nurses.

DETAILED DESCRIPTION:
Allocation of the nurses to the procedure groups (with VR-G and no VR-G procedures) is done with using Random Allocation Software program.

Among the with VR-G procedure:

The nurses were asked to watch a relaxing video with using VR-G for 20 minutes at their break time. The researcher visited the nurses at the beginning of the working shift and asked the nurse stress scale items to them in the nursing room, scheduled a break period with them individually and visited them again at the scheduled time. Then, the researcher prepared the video and googles, asked nurses to sit on the chair in the nursing room at the surgical unit, helped them to wear the VR-G and let them alone to watch the video for 20 minutes.

At the end of their working shift, the researcher visited them and asked the scale items once again.

Among the no VR-G procedure:

The nurses did not watch any video and copleted their routine working shift and break times. The researcher visited the nurses at the beginning and at the end of their working shift and asked the nurse stress scale items to them in the nursing room.

ELIGIBILITY:
Inclusion Criteria:

* working in a surgical unit for at least one year
* able to use virtual reality glasses
* volunteering to participate in this study

Exclusion Criteria:

* having a visual and/or audial problems
* leaving surgical unit for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-01-24 (Actual); Primary Completion 2023-07-24 (Actual); Study Completion 2023-08-04 (Actual)

PRIMARY OUTCOMES:
Stress level | At the beginning and end of nurses daily working shift through study completion, an average of six months.
  will be evaluated with using the "Nurse Stress Scale (NSS)" which is developed by Gray-Toft and Anderson and, translated and validated in Turkish by Mert, Sayilan and Baydemir. This scale consists of seven subcategories and 34 positive items rated using a 4-point Likert scoring system "1-never", "2-sometimes", 3-often," "4-very often". The total scale score, which reflects the frequency of the stress experienced by nurses, ranges from 34 to 136 points. A higher score indicates more frequent stress, while a lower score indicates less stress for the same situations.

CONTACTS AND LOCATIONS:
Overall Officials: Seher Ünver, Principal Investigator — Trakya University; Seda C Yeniğün, Principal Investigator — Akdeniz University
Locations (2):
- Turkey (Türkiye) (2):
  - Trakya University, Edirne, Turkey
  - Seher Ünver, Edirne

IPD SHARING:
Plan to Share IPD: No